CLINICAL TRIAL: NCT06777823
Title: Rejection Sensitivity and Puberty in Mental Health Vulnerability to Social Media Experiences in Early Adolescent Girls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis University (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01MH135480-01A1 (NIH)
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Rejection Sensitivity; Puberty; Psychopathology
Keywords: puberty; rejection sensitivity; psychopathology; social media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants complete the study intervention
  Interventions: Behavioral: Social Rejection Task

INTERVENTIONS:
Behavioral: Social Rejection Task — All participants will receive this

SUMMARY:
This longitudinal study is designed to test bidirectional relationships between preteen girls' mental health and social media experiences. We will explore how pubertal development and experiences of rejection influence these relationships.

ELIGIBILITY:
Inclusion Criteria:

* female aged 10-11 years
* engagement in social media use
* proficient in the English language
* family/personal device that can complete daily diaries

Exclusion Criteria:

* previously diagnosed chronic medical illness
* autism spectrum disorder
* significant developmental or speech delay
* endocrine disorder
* not assigned female at birth (AFAB)

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychopathology symptoms parent report | "Through study completion, an average of two years"
  Measured via the KSADS interview
Psychopathology symptoms child report | "Through study completion, an average of two years"
  Measured via the KSADS interview
Daily Diary Social Media experiences | Through study completion, an average of two years
  Assessed through daily diary reports (e.g., 'Did you use social media today?")
MicroEMA Social Media experiences | Through study completion, an average of two years
  Assessed through microEMA prompt (e.g., 'using Social Media?")
Social Media experiences child report | Through study completion, an average of two years
  Assessed through a screen time questionnaire
Social Media experiences parent report | Through study completion, an average of two years
  Assessed through a screen time questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes